CLINICAL TRIAL: NCT01694823
Title: A Prospective Open-label Multi-center Study to Demonstrate the Safety and Efficacy of Cells Sheet-Autologous Chondrocyte Implantation（CS-ACI）for the Treatment of Articular Cartilage Defects
Brief Title: Safety and Efficacy Study of Cells Sheet-Autologous Chondrocyte Implantation to Treat Articular Cartilage Defects
Acronym: CS-ACI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yan Jin (Other)
Collaborators: Xijing Hospital (Other); Tang-Du Hospital (Other)
Responsible Party: Sponsor-Investigator, Yan Jin, Director of Research and Development Center for Tissue Engineering, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-ACI2012001
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Osteochondritis; Osteochondritis Dissecans; Joint Diseases
Keywords: Cartilage repair; Cartilage defects; cell sheet; Autologous chondrocyte implantation
MeSH Terms: conditions — Osteochondritis; Osteochondritis Dissecans; Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CS-ACI (Experimental): Group/Cohort Label： pretherapy post-treatment
  Group/Cohort Description ：The CS-ACI is used to prepare cell sheet and implant to the Cartilage defects.The arm of safety and efficacy are compared preoperative observation with postoperative observation.
  Interventions: Drug: CS-ACI

INTERVENTIONS:
Drug: CS-ACI — Procedure: Self-control. Cells Sheet-Autologous Chondrocyte Implantation(CS-ACI) includes an arthroscopy for harvesting of cartilage 6-8 weeks prior to the open cartilage surgery. Other Names:
  Cells Sheet-Autologous Chondrocyte Implantation （CS-ACI）
  Other Names: Cells Sheet-Autologous Chondrocyte Implantation（ CS-ACI）

SUMMARY:
In this study,the Autologous chondrocyte implantation (ACI)technology and cell sheet technology are used to Cells Sheet-Autologous Chondrocyte Implantation(CS-ACI) for treating Cartilage Defects.The Safety and Efficacy Study of CS-ACI are evaluated.

DETAILED DESCRIPTION:
All procedures are carried out after obtaining informed written consent from patients. Cartilage tissue is acquired from the Non-weight-bearing area of patients. chondrocyte are isolated and grown in culture for 6-8 weeks. After this time interval, the cells are reprocessed and the cell sheet is obtained. Implantation of the chondrocyte sheet into the Cartilage defect of the keen.The patients will be assessed clinically with scoring systems preoperatively as well as 24 months postoperatively to assess relief of symptoms and joint function. Radiological assessment (MRIs)of the affected joints will be performed at the same time points aforementioned to assess integrity of the formed cartilage. Second look arthroscopy and biopsy will also be performed to histologically assess the repair tissue and grade it via arthroscopic grading system according to the International Cartilage Repair Society guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age: between 18 and 50 years
* Defect: isolated ICRS grade III or IV single defect chondral lesions on Articular Cartilage
* Defect size: 2.5 to < 5 cm2 after debridement to healthy cartilage up to 6 mm in depth.
* Nearly intact chondral structure surrounding the defect as well as an intact corresponding joint area
* Informed consent signed and dated by patient and Patient understands the strict rehabilitation protocol and follow-up programme and is willing to follow it
* No ligament damage or ligament damage after reconstruction

Exclusion Criteria:

* Patients younger than 18 years and older than 50 years.
* Arthrofibrosis or Ankylosis
* Arthritis
* Obesity
* Infectious diseases
* the other cases of patients which Doctors determine not participate in the trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-07 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in the MRI | 3month,6 month, 12 months, 24 months

SECONDARY OUTCOMES:
Change from Baseline in the Lysholm | 3month,6 month, 12 months, 24 months
Change from Baseline in the Knee injury and Osteoarthritis Outcome Score (KOOS)Which consists of five sub- categories = Pain, ADL, QOL, Symptoms, Sport | 3month,6 month, 12 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yan, Ph.D, Study Director — Research and Development Center for Tissue Engineering,Fourth Military Medical University
Locations (3):
- China (3):
  - Xijing Hospital, Xi'an
  - Tangdu Hospital, Xi'an
  - Xi'An Honghui Hospital, Xi'an

REFERENCES:
- [Background] Ebihara G, Sato M, Yamato M, Mitani G, Kutsuna T, Nagai T, Ito S, Ukai T, Kobayashi M, Kokubo M, Okano T, Mochida J. Cartilage repair in transplanted scaffold-free chondrocyte sheets using a minipig model. Biomaterials. 2012 May;33(15):3846-51. doi: 10.1016/j.biomaterials.2012.01.056. Epub 2012 Feb 25. PMID 22369960